CLINICAL TRIAL: NCT04478357
Title: AN OPEN-LABEL, RANDOMIZED, SINGLE-DOSE, 4 PERIOD, 4 TREATMENT, 2 SEQUENCE, TWO 2 WAY CROSSOVER, BIOEQUIVALENCE STUDY IN HEALTHY PARTICIPANTS COMPARING 4 MG AND 8 MG FESOTERODINE EXTENDED RELEASE TABLETS (TOVIAZ(TM)), MANUFACTURED AT ZWICKAU VERSUS FREIBURG
Brief Title: BIOEQUIVALENCE STUDY IN HEALTHY PARTICIPANTS COMPARING 4 MG AND 8 MG FESOTERODINE EXTENDED-RELEASE TABLETS (TOVIAZ™), MANUFACTURED AT ZWICKAU VERSUS FREIBURG
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: A0221106; 2014-002783-32 (EudraCT Number)
Record Dates: First submitted 2020-07-01; First posted 2020-07-20 (Actual); Last update posted 2021-05-07 (Actual); Status verified 2021-05

CONDITIONS: Neurogenic Detrusor Overactivity
Keywords: Phase I; Fesoterodine beads- in-capsule; bioequivalence; Pharmacokinetics; Toviaz

STUDY DESIGN:
Intervention Model Description: This is an open-label, randomized, single-dose, 4-period, 4-treatment, 2-sequence, two 2-way crossover study in healthy participants. This study will assess the BE of Fesoterodine (Toviaz™) 4 mg and 8 mg ER tablets manufactured at Zwickau (Reference) versus Freiburg (Test). Study participants will include healthy male and/or female individuals between the ages of 18 and 55 years, inclusive. Approximately 18 participants who fulfill entry criteria will be randomized to 1 of the 2 treatment sequences as shown in the table below.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Treatment A (Other): 4 mg fesoterodine ER tablet manufactured at Zwickau.
  Interventions: Drug: 4 mg Fesoterodine ER tablet from Zwickau
- Treatment B (Other): 4 mg fesoterodine ER tablet manufactured at Freiburg
  Interventions: Drug: 4 mg fesoterodine ER tablet from Freiburg
- Treatment C (Other): 8 mg fesoterodine ER tablet manufactured at Zwickau
  Interventions: Drug: 8 mg fesoterodine ER tablet from Zwickau
- Treatment D (Other): 8 mg fesoterodine ER tablet manufactured at Freiburg.
  Interventions: Drug: 8 mg fesoterodine ER tablet from Freiburg

INTERVENTIONS:
Drug: 4 mg Fesoterodine ER tablet from Zwickau — Manufactured at Zwickau
  Arms: Treatment A
Drug: 4 mg fesoterodine ER tablet from Freiburg — Manufactured at Freiburg
  Arms: Treatment B
Drug: 8 mg fesoterodine ER tablet from Zwickau — Manufactured at Zwickau
  Arms: Treatment C
Drug: 8 mg fesoterodine ER tablet from Freiburg — Manufactured at Freiburg
  Arms: Treatment D

SUMMARY:
Fesoterodine (Toviaz™) extended-release (ER) tablets are currently manufactured by Aesica Pharmaceuticals, Zwickau, Germany (Zwickau). An additional manufacturing location at Pfizer Freiburg, Germany (Freiburg) has been identified. This pivotal bioequivalence (BE) study is being conducted to satisfy the United States (US) Food and Drug Administration (FDA) regulatory requirements for the qualification of the Freiburg manufacturing site.

Overall Study Design This is an open-label, randomized, single-dose, 4-period, 4-treatment, 2-sequence, two 2-way crossover study in healthy participants. This study will assess the BE of Fesoterodine (Toviaz™) 4 mg and 8 mg ER tablets manufactured at Zwickau (Reference) versus Freiburg (Test). Study participants will include healthy male and/or female individuals between the ages of 18 and 55 years, inclusive. Approximately 18 participants who fulfill entry criteria will be randomized to 1 of the 2 treatment sequences as shown in the table below.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female participants must be 18 to 55 years of age, inclusive, at the time of signing the informed consent document (ICD).
2. Male and female participants who are overtly healthy as determined by medical evaluation including a detailed medical history, complete physical examination, cardiovascular tests including blood pressure (BP), pulse rate measurement and 12-lead ECG, and clinical laboratory tests.
3. Participants who are willing and able to comply with all scheduled visits, treatment plan, laboratory tests, lifestyle considerations, and other study procedures.
4. Body mass index (BMI) of 17.5 to 30.5 kg/m2; and a total body weight >50 kg (110 lb).
5. Capable of giving signed informed consent as described in Appendix 1, which includes compliance with the requirements and restrictions listed in the informed consent document (ICD) and in this protocol.

Exclusion Criteria

1. Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurological, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing).
2. Any condition possibly affecting drug absorption (eg, gastrectomy).
3. History of human immunodeficiency virus (HIV) infection, hepatitis B, or hepatitis C infection; positive testing for HIV, hepatitis B surface antigen (HBsAg), or hepatitis C antibody (HCVAb). Hepatitis B vaccination is allowed.
4. Other acute or chronic medical or psychiatric condition including recent (within the past year) or active suicidal ideation or behavior or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the participant inappropriate for entry into this study.
5. History of allergy or hypersensitivity to fesoterodine fumarate or tolterodine tartrate, soya, or any of the excipients in the investigational drug product.
6. History of uncontrolled narrow angle glaucoma, myasthenia gravis, gastric retention, severe ulcerative colitis and toxic megacolon.
7. Evidence or history of clinically significant urologic disease, urinary retention, obstructive disturbance of bladder emptying, micturition disturbance, nocturia or pollacisuria (eg, benign prostate hyperplasia, urethral stricture, recurrent urinary tract infections).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2019-11-12 (Actual); Primary Completion 2020-11-12 (Actual); Study Completion 2020-11-12 (Actual)

PRIMARY OUTCOMES:
Cmax | 0, 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 24, 30, 36, and 48 hours
  Maximum Observed Plasma Concentration (Cmax) of 5-Hydroxymethyl-tolterodine (5-HMT)
AUCinf (if data permit, otherwise AUClast) | 0, 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 24, 30, 36, and 48 hours
  Area Under the Curve From Time Zero to Extrapolated Infinite Time [AUC (0 - ∞)] of 5-Hydroxymethyl-tolterodine (5-HMT)

SECONDARY OUTCOMES:
AUCLast | 0, 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 24, 30, 36, and 48 hours
  Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) of 5-Hydroxymethyl-tolterodine (5-HMT)
Tmax | 0, 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 24, 30, 36, and 48 hours
  Time to Reach Maximum Observed Plasma Concentration (Tmax) of 5-Hydroxymethyl-tolterodine (5-HMT)
t1/2 | 0, 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 24, 30, 36, and 48 hours
  Plasma Decay Half-Life (t1/2) of 5-Hydroxymethyl-tolterodine (5-HMT)
Number of Participants With Treatment Emergent Treatment-Related Adverse Events (AEs) | Day -28 to day -1, 0, 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 24, 30, 36, and 48 hours, Day 28 to 35 and on early termination
Number of Participants With Clinically Significant Change From Baseline in Vital Signs | Day -28 to day -1, 0, 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 24, 30, 36, and 48 hours, Day 28 to 35 and on early termination
Number of Participants With Clinically Significant Change From Baseline in Laboratory Abnormalities | During screening

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Brussels Clinical Research Unit, Brussels, Bruxelles-capitale, Région de, Belgium

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=A0221106